CLINICAL TRIAL: NCT02717273
Title: A Randomized, Prospective Study of Surgical Site Infections in Liver Transplant Patients Receiving Three Days of Peri-operative Antibiotic Prophylaxis Versus Intra-operative Antibiotics Only
Brief Title: Surgical Site Infections After Liver Transplantation Based on Perioperative Antibiotics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Robert Sawyer, MD, Profesor of Surgery, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-HSR#14971; T32AI078875 (NIH)
Record Dates: First submitted 2016-03-02; First posted 2016-03-23 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Liver Transplantation; Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Anti-Bacterial Agents; Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard peri-operative antibiotics (Active Comparator): The standard of care at the University of Virginia Medical Center for liver transplantation patients is a 3.375 gram dose of piperacillin / tazobactam (Zosyn®) at the time of induction of anesthesia, though this dose may be adjusted for renal insufficiency. This dose is repeated during the operation every six hours.
  Interventions: Drug: standard; Other: liver transplant
- extended three-day course of antibiotics (Experimental): For those patients randomized to the study group, antibiotics will be started as per the usual intra-operative dosing regimen, then continued to provide coverage for 72 hours.
  This is typically provided as additional doses of 3.375 grams of piperacillin / tazobactam (Zosyn®) every 8 hours for 3 total days (giving a total of 72 hours of antibiotic coverage), though this may be altered based on kidney function.
  Interventions: Drug: extended; Other: liver transplant

INTERVENTIONS:
Drug: standard — peri-operative antibiotic regimen only
  Other Names: Peri-operative only antibiotics
  Arms: standard peri-operative antibiotics
Drug: extended — extended three-day course of antibiotics
  Other Names: Extended, three-day antibiotics
  Arms: extended three-day course of antibiotics
Other: liver transplant — orthotopic liver transplantation

SUMMARY:
This study will be to prospectively determine differences in Surgical Site Infection (SSI) if a prolonged course of post-operative antibiotics are used following liver transplantation.

DETAILED DESCRIPTION:
This study will be to prospectively determine differences in SSI if a prolonged course of post-operative antibiotics are used following liver transplantation. All adult patients, admitted to the University of Virginia (UVA) Medical Center for first-time liver transplantation will be randomized to the standard of care of peri-operative antibiotics or extended course of three total days.

Patients will be evaluated primarily for the presence of post-operative surgical site infections but also for fever, elevated white blood counts, secondary infections (urinary tract, pneumonia, and blood stream), length of hospital stay, graft loss, and mortality for 30 days after liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years of age.
* Eligible for liver transplantation by UVA standard protocol.
* First-time transplantation.
* No active infections - requiring antibiotics - excluding antifungals.

Exclusion Criteria:

* All patients < 18 years of age.
* Previous liver transplantation.
* Active infections - requiring antibiotics.
* Allergy to all standard peri-operative antibiotics (piperacillin/tazobactam or UVA standard alternatives for Penicillin allergic patients: ciprofloxacin and vancomycin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Sawyer, MD, Principal Investigator — UVA

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chan S, Ng S, Chan HP, Pascoe EM, Playford EG, Wong G, Chapman JR, Lim WH, Francis RS, Isbel NM, Campbell SB, Hawley CM, Johnson DW. Perioperative antibiotics for preventing post-surgical site infections in solid organ transplant recipients. Cochrane Database Syst Rev. 2020 Aug 4;8(8):CD013209. doi: 10.1002/14651858.CD013209.pub2. PMID 32799356

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Peri-operative Antibiotic Regimen: The standard of care at the University of Virginia Medical Center for liver transplantation patients is a 3.375 gram dose of piperacillin / tazobactam (Zosyn®) at the time of induction of anesthesia, though this dose may be adjusted for renal insufficiency. This dose is repeated during the operation every six hours.
  standard: peri-operative antibiotic regimen only
  steroids: 500mg methylprednisolone intravenously
  liver transplant: orthotopic liver transplantation
- Extended Three-day Course of Antibiotics: For those patients randomized to the study group, antibiotics will be started as per the usual intra-operative dosing regimen, then continued to provide coverage for 72 hours.
  This is typically provided as additional doses of 3.375 grams of piperacillin / tazobactam (Zosyn®) every 8 hours for 3 total days (giving a total of 72 hours of antibiotic coverage), though this may be altered based on kidney function.
  extended: extended three-day course of antibiotics
  steroids: 500mg methylprednisolone intravenously
  liver transplant: orthotopic liver transplantation
Period: Overall Study
Arm/Group | Standard Peri-operative Antibiotic Regimen | Extended Three-day Course of Antibiotics
Started | 52 | 50
Completed | 49 | 48
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Peri-operative Antibiotic Regimen | Extended Three-day Course of Antibiotics | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 44 | 90
  >=65 years | 6 | 6 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [51 to 58] | 58.5 [55 to 61] | 57.5 [52 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 11 | 33
  Male | 30 | 39 | 69
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 50 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Development of Surgical Site Infections
Description: development of surgical site infection, including superficial and deep incisional and organ space surgical site infections
Time Frame: within 30 days from surgery
Population: Had liver transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Peri-operative Antibiotic Regimen | Extended Three-day Course of Antibiotics
Number analyzed (Participants) | 48 | 49
Participants | 9 | 13

2. Secondary Outcome: Number of Subjects With Post-operative Fever
Description: fever above 38.5 degrees Celsius 24 hours after the end of the liver transplant
Time Frame: 24 hours from surgery
Population: Had liver transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Peri-operative Antibiotic Regimen | Extended Three-day Course of Antibiotics
Number analyzed (Participants) | 48 | 49
Participants | 6 | 7

3. Secondary Outcome: Number of Subjects With Elevated White Blood Count (WBC)
Description: above 15,000 within 24hours after the end of the liver transplant
Time Frame: 24 hours from surgery
Population: Had liver transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Peri-operative Antibiotic Regimen | Extended Three-day Course of Antibiotics
Number analyzed (Participants) | 48 | 49
Participants | 42 | 41

4. Secondary Outcome: Number of Subjects With Nosocomial Infection
Description: diagnosis of any new infection other than an SSI within 30 days from surgery
Time Frame: within 30 days from surgery
Population: Had liver transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Peri-operative Antibiotic Regimen | Extended Three-day Course of Antibiotics
Number analyzed (Participants) | 48 | 49
Participants | 8 | 11

5. Secondary Outcome: Length of Hospital Stay
Description: days hospitalized after liver transplant
Time Frame: within 30 days from surgery
Population: Had liver transplant
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard Peri-operative Antibiotic Regimen | Extended Three-day Course of Antibiotics
Number analyzed (Participants) | 48 | 49
days | 7.5 [6.5 to 11] | 7.5 [6 to 12]

6. Secondary Outcome: Number of Subjects With Graft Loss
Description: complete loss of liver function in recipient
Time Frame: within 30 days from surgery
Population: Had liver transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Peri-operative Antibiotic Regimen | Extended Three-day Course of Antibiotics
Number analyzed (Participants) | 48 | 49
Participants | 7 | 6

7. Secondary Outcome: Number of Subjects With Mortality
Description: death within 30 days of liver transplant
Time Frame: within 30 days from surgery
Population: Had liver transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Peri-operative Antibiotic Regimen | Extended Three-day Course of Antibiotics
Number analyzed (Participants) | 48 | 49
Participants | 1 | 1

ADVERSE EVENTS:
Arm/Group | Standard Peri-operative Antibiotic Regimen | Extended Three-day Course of Antibiotics
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/49
Other Adverse Events (participants affected / at risk) | 0/48 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes